CLINICAL TRIAL: NCT03315468
Title: French National Cohort of Patients With Melanoma (Any Stage). Network for Research and Clinical Investigation, the RIC-Mel Network.
Brief Title: French Clinical Datbase of Melanoma Patients (RIC-Mel)
Acronym: RIC-Mel
Status: Recruiting | Type: Observational
Sponsor: Nantes University Hospital (Other)
Collaborators: CENGEPS (Unknown); Bristol-Myers Squibb (Industry); Hoffmann-La Roche (Industry); GlaxoSmithKline (Industry); Amgen (Industry)
Responsible Party: Sponsor
Other Study IDs: Prog 09/37-11
Record Dates: First submitted 2017-10-06; First posted 2017-10-20 (Actual); Last update posted 2025-07-22 (Actual); Status verified 2025-07

CONDITIONS: Melanoma (Skin)
Keywords: melanoma; database; cohort
MeSH Terms: conditions — Melanoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
With a high incidence, low survival rates and limiter availability of effective treatment, melanoma is one of the research priorities for health authorities. Optimizing the development of both academic and private research requires the availability information on the features of patients.

To meet this need, the French Multidisciplinary Melanoma Group (GMFMel) in collaboration with INCa (French National Cancer Institute), the CeNGEPS (National Centre for Healthcare Products Trial Management) and the CIC-BT0503 from Nantes University Hospital (Biotherapy Clinical Centre of Investigation) has set up in April 2011 a Clinical Investigation Network for melanoma, called the CeNGEPS-GMFMel network. Nowadays, the network is named :

RIC-Mel : network for Research and Clinical Investigation on Melanoma. Aims of the network are to promote translational and epidemiological projects as well as to optimize the achievements of clinical trials.

To achieve these goals, a database was launched in 2012 that gives a permanently updates mapping of melanoma treated in France with the key information needed for any research projects.

DETAILED DESCRIPTION:
The RIC-Mel network federate clinicians researchers working in clinical and translational research for melanoma and carrying out patients inclusions in the clinical trials. These clinicians are working on clinical cancerology and dermatology sites located throughout the French national territory. Nowadays, the RIC-Mel network consists of 49 centers: 43 public dermatology centers (Hospital centers) and 6 private centers (Cancer centers). The RIC-Mel network is coordinated by Pr B. DRENO (Nantes University Hospital) and Pr C. LEBBE (Saint-Louis Hospital, AP-HP, Paris).

The RIC-Mel database is referred as one of the privileged access to any research program on melanoma by the Cancerology Group of the French Society of Dermatology.

The RIC-Mel database has been approved by French health authorities, both ethically and for confidentiality of data (CCTIRS and CNIL). The database is available on the internet at any given moment thanks to a secure connection. All data are treated confidentially. The active file of patients with melanoma from each participating center is available in the database. All patients agreed to participate may be included in the database, regardless of their stage. Clinical data are collected thanks two forms :

* Part I key clinical data for any clinical trial Primary tumour (date of surgery, breslow…), lymph node removal (date, number of invaded lymph node…), AJCC stage, Mutation status, melanoma antigens, melanoma treatments (type, dates) and death.
* Part II: additional data for epidemiological and translational research Family history of melanoma, metastases (type, date of diagnosis…), HLA A and B type, additional information on treatments (dose, overall response, grade 3 or 4 side effects with the type, action on treatment and outcome).

In September 2017, more than 20,000 patients with melanoma had been included in the RIC-Mel database, with the following distribution: around 75% of primary stages (0 to II) and 25 % of metastatic stages (III and IV).

ELIGIBILITY:
Inclusion Criteria:

* Patient with melanoma, of any stage,
* Patient agreed to participate.

Exclusion Criteria:

* Individuals under court protection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with melanoma
Sampling Method: Non-Probability Sample
Enrollment: 16000 (Estimated)
Dates: Start 2012-03-01 (Actual); Primary Completion 2030-03-01 (Estimated); Study Completion 2030-03-01 (Estimated)

PRIMARY OUTCOMES:
Overall survival of melanoma patients included in the RIC-Mel database | 5 years
  Overall survival if defined as the time between the primary melanoma tumour removal and the death or the date of data extraction from the RIC-Mel database for alive patients.

SECONDARY OUTCOMES:
Percentage of melanoma patients included in the RIC-Mel database categorized by genders | through study completion, an average of 5 years
  Distribution of females and males
Percentage of melanoma patients included in the RIC-Mel database categorized by histological subtypes | Day 1
  Histological subtypes of primary melanoma were categorized as Superficial spreading melanoma, nodular, lentigo maligna melanoma, acral lentiginous melanoma, mucosal, ocular, unknown primary melanoma, and others subtypes. This information is collected from medical records of each patient
Percentage of melanoma patients included in the RIC-Mel database categorized by breslow thickness | day 1
  Breslow thickness is defined as the total vertical height of the melanoma, from the very top (called the granular layer) to the area of deepest penetration in the skin. Breslow thickness is the one of the important prognostic factor and it is commonly reported that the higher the Breslow thickness, the worse the prognosis. This information is collected from medical records of each patient. The classifications were lesser than or equal to (≤) 1.0 millimeters (mm), 1.01 - 2.0 mm, 2.01 - 4.0 mm, greater than (>) 4.0 mm and Unknown.
Percentage of melanoma patients included in the RIC-Mel database categorized by ulceration | day 1
  Ulceration is defined as an erosion of the first primary tumour, associated with the death of cancer cells in the tumour center. Ulceration is, with breslow thickness, another important prognostic factor. Ulceration is associated with a worth prognostic. This information is collected from medical records of each patient. The classifications were Yes, No and Unknown.
Percentage of melanoma patients included in the RIC-Mel database categorized by Melanoma stage | day 1
  Melanoma stages were categorized (according to American Joint Committee on Cancer [AJCC]) as 0 (in situ melanoma), I and II (only primary tumour without any metastasis), III (locally advanced stage of melanoma regarding location of the primary tumour with lymph nodes and/or cutaneous metastasis), IV (advanced stage of melanoma with lymph nodes and/or cutaneous distant metastasis or any other type of metastasis). This information is collected from medical records of each patient
Percentage of Participants With Mutation Status | Day 1
  Presence or absence of mutations in the BRAF, NRAS and ckit oncogenes were determined thanks to each's centres practices. This information is collected from medical records of each patient.The classifications for each gene were Yes (mutated), No (non-mutated = wild type) and Unknown (no research).
Percentage of treatment types among melanoma stage | through study completion, an average of 5 years
  Possible treatments types: Radiotherapy, Immunotherapy, Targeted therapies, Chemotherapy, Experimental treatment, Interferon, Others (for surgical approaches). All treatments reported in the RIC-Mel database only concerned those provided in the care of melanoma. This information is collected from medical records of each patient.
Progression-free survival of melanoma patients included in the RIC-Mel database | 5 years
  Progression-free survival if defined as the time between the primary melanoma tumour removal and the appearance of the first metastasis.

CONTACTS AND LOCATIONS:
Overall Officials: Gaëlle Quereux, PU-PH, Principal Investigator — Nantes University Hospital
Locations (1):
- Nantes University Hospital, Nantes, France